CLINICAL TRIAL: NCT05858879
Title: Notification of Incidental Coronary Artery Calcium in Patients With Atherosclerotic Cardiovascular Disease (NOTIFY-ASCVD)
Acronym: NOTIFY-ASCVD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Fatima Rodriguez, Associate Professor of Medicine (Cardiovascular Medicine), Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 70362
Record Dates: First submitted 2023-05-05; First posted 2023-05-15 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: ASCVD; Coronary Artery Calcification

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized to: 1) notification of presence of CAC with a CT scan image; 2) notification of presence of CAC without a CT scan image; 3) or usual care.
Who Masked: Participant, Care Provider
Masking Description: In the usual care arm, patients or clinicians will not be notified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Notification with a CAC image (Experimental): Notification of presence of CAC with a CT scan image and the ACC/AHA guideline recommendation for initiation of lipid-lowering therapy.
  Interventions: Other: Notification of patients and clinicians
- Notification without a CAC image (Experimental): Notification of presence of CAC without a CT scan image and the ACC/AHA guideline recommendation for initiation of lipid-lowering therapy.
  Interventions: Other: Notification of patients and clinicians
- Usual care (No Intervention): The usual care arm will not receive any additional notification beyond the standard of care. If the intervention is successful, we will notify patients in the usual care arm of the presence of CAC and the ACC/AHA guideline recommendation for initiation of lipid-lowering therapy.

INTERVENTIONS:
Other: Notification of patients and clinicians — Notification Patients randomized to notification will receive a message sent by either the electronic health record (EHR) patient portal or US mail that will inform them of the CAC identified on their previous chest CT scan (with or without an image) and a recommendation that they discuss this finding and initiation of lipid-lowering therapy with their clinician. The clinicians will be notified of these findings by an earlier EHR message that will be sent 2 weeks before the patient notification.
  Two months after the initial notification, patients and their clinicians who are randomized to notification arms will receive a second message similar to the initial notification.
  Arms: Notification with a CAC image; Notification without a CAC image

SUMMARY:
Estimate the impact of notifying both patients and their clinicians of the presence of incidental coronary artery calcium (CAC) on initiation of lipid-lowering therapy in patients with ASCVD who are not receiving lipid-lowering therapy.

DETAILED DESCRIPTION:
This is a randomized quality improvement (QI) project evaluating the impact of notifying patients and their clinicians (primary care, cardiologists, neurologists, or vascular surgeon) of incidental CAC detected on a prior chest CT scan. Patients will be identified by screening previous non-gated chest CT scans and electronic health records. The presence of CAC will be confirmed by a radiologist. Eligible patients will be randomized to: 1) notification of presence of CAC with a CT scan image; 2) notification of presence of CAC without a CT scan image; 3) or usual care.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of CAC on non-gated chest CT scans performed from 2021 to 2025
2. Age <85 years
3. Diagnosis of ASCVD(coronary artery disease, peripheral artery disease, or cerebrovascular disease)
4. Visit to Stanford affiliated clinician since 2022 at one of the following Stanford clinics including University affiliated clinics:

   1. Internal Medicine
   2. Family Medicine
   3. Cardiology
   4. Neurology
   5. Vascular surgery
5. Primary language is English or Spanish

Exclusion Criteria:

1. No diagnosis of ASCVD
2. Patients receiving lipid-lowering therapy
3. Dementia
4. Metastatic cancer or active cancer undergoing chemotherapy
5. Hospice

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Initiation of lipid-lowering therapy | Month 6
  Number of patients who had initiation of lipid-lowering therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No